CLINICAL TRIAL: NCT04123587
Title: Genetic Variants Replication Study Associated With Dependence on Sulfonylurea in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hye Seung Jung, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU
Record Dates: First submitted 2019-09-10; First posted 2019-10-11 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus
Keywords: Sulfonylurea
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sulfonylurea-dependent (Experimental): Sulfonylurea is replaced by alternative oral hypoglycemic agent.
  Interventions: Drug: discontinuation of Sulfonylureas

INTERVENTIONS:
Drug: discontinuation of Sulfonylureas — 1. Discontinuation of sulfonylurea, alternative drug administration.
  2. If there is a significant increase in blood glucose, it is considered as a sulfonylurea-dependent patient. Discontinue the alternative drug and resume the sulfonylurea, and monitor for 12 weeks or until stabilization of blood glucose at short intervals.
  3. if blood glucose levels are within optimal range after replacement of sulfonylureas with other agents, the patient is regard as non-SU-dependent
  Other Names: other oral anti-diabetics instead of sulfonylureas

SUMMARY:
This study was designed to reproduce candidate single nucleotide variants found by whole exome sequencing in some type 2 diabetic patients dependent on sulfonylurea in a separate patient group. The validation of the dependence-related variations performed in this study is expected to help decision-making in the clinical use of sulfonylurea in the future.

DETAILED DESCRIPTION:
Sulfonylurea, one of the oral hypoglycemic agents, is the oldest and most widely used drug. The use of sulfonylurea was overwhelming compared to metformin especially in East Asia, where insulin secretion was notable during the pathophysiology of type 2 diabetes. However, sulfonylurea causes hypoglycemia and weight gain, increases cardiovascular disease and mortality compared to other oral preparations. With the recent development of other oral hypoglycemic agents for lowering blood glucose without the risk of hypoglycemia and with cardiovascular protection, sulfonylurea is in a decreasing state of use worldwide.

But some patients tend to be highly dependent on sulfonylurea for blood glucose control. It suggests that there will be a group of patients whose the action of sulfonylurea is strongly influenced by genetic factor, since insulin secretion of pancreatic beta cells is very hereditary, genetic variations that increase the risk of type 2 diabetes are found mainly in genes related to beta cell dysfunction rather than insulin resistance, and the more risk variants of type 2 diabetes, the less likely the effect of sulfonylurea is.

The investigators had performed whole exome sequencing in patients showing dependence on sulfonylurea and identified tens of candidate variants.

In this study, the investigators will select patients with dependence on sulfonylurea by prospective intervention (by discontinuing and resuming sulfonylurea) and perform genetic tests.

ELIGIBILITY:
Inclusion Criteria:

Among patients with type 2 diabetes who visited Seoul National University Hospital endocrinology outpatient clinic, all of criteria (1)-(4) are satisfied

1. Adults over 19 years
2. More than 10 years of diabetes
3. Low dose sulfonylurea use: Equivalent capacity 2 mg or less of glimepiride
4. Less than 7.5% of glycated hemoglobin for more than 6 months
5. estimated glomerular filtration rate > 50 mL/min/1.73㎡

Exclusion Criteria:

* Type 1 diabetics
* Insulin user
* Patients diagnosed with cardiovascular disease, cancer, and other critical illness within 6 months before the study
* Patients with severe hypertension
* Patients with treatment or diseases that may have a significant effect on blood glucose levels, such as glucocorticoids and thyrotoxicosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
the list of previously found candidate variants which are observed in the slufonylurea-dependent patients but not in the non-dependent patients | 20 weeks
  Dependency on sulfonylurea-dependency is determined according to changes in HbA1c by use of sulfonylurea. The 'previously found candidate variants' are the results from whole exome sequencing in patients showing dependence on sulfonylurea as a screening before.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Seung Jung, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea